CLINICAL TRIAL: NCT02120001
Title: Silver-coated Endotracheal Tube Cleaned With a Novel Mechanism for Secretion Removal: a Randomized Controlled Clinical Study.
Brief Title: Efficacy Study on Silver-coated ETT Cleaned With a Novel Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Anesthesia and Critical Care MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DAN1000AM
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Ventilator Associated Pneumonia; Critically Ill
Keywords: Medical Devices; Ventilator-Associated Pneumonia (VAP); Ventilator-Associated Events (VAE); Endotracheal Tube; Microbial Diversity; Drug-Resistance; biofilms; endotracheal intubation; mechanical ventilation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETT cleaning maneuver (Experimental): Patients randomized to the treatment group will undergo an ETT cleaning maneuver with endOclear three times a day (every 8 hours) for the whole intubation period in addition to the standard of care.
  Interventions: Device: ETT cleaning maneuver
- Standard of care (No Intervention): In the protocol no intervention is planned for the control group, which will therefore be treated with blind suctioning as per caregiver clinical decision.

INTERVENTIONS:
Device: ETT cleaning maneuver — EndOclear is a commercially available device. It consists of an endotracheal tube cleaning apparatus with a flexible central tube and a cleaning device at its distal end. In operation, the collapsed cleaning apparatus is inserted into the ETT through a Y-shaped connector. The device is then expanded by a safety toggle protected trigger mechanism that, when fired, presses the device's smooth silicone disc against the inside surface of the endotracheal tube. The cleaning apparatus is then pulled out of the endotracheal tube removing mucus deposits and secretions.
  We plan to add the use of endOclear to the standard ICU practice, scheduling the systematic use of the device every 8 hours for the whole intubation period.
  Other Names: endOclear
  Arms: ETT cleaning maneuver

SUMMARY:
The purpose of this study is to test the efficacy of a novel cleaning device in keeping silver-coated endotracheal tubes free from bacterial colonization.

DETAILED DESCRIPTION:
Several studies have suggested that biofilm formation inside the ETT plays a pivotal role in VAP development and drug-resistance induction. Silver-coated ETT have proven effective in delaying but not in preventing ETT colonization and biofilm formation, due to a barrier effect of biofilm and accumulated debris. Advanced ETT cleaning devices are able to remove debris and biofilm and reduce the total ETT microbial load to a certain extent. The Investigators hypothesize that the routine use of endOclear in patients intubated with a silver-coated ETT will reduce ETT microbial colonization. The Investigators therefore want to assess the reduction of ETT microbial colonization in patients intubated with a silver-coated ETT and cleaned with endOclear compared to the current standard of care of silver-coated ETT (blind suctioning). They plan to achieve this result by analyzing the tubes of each enrolled patient after it has been removed, either because the patient does not need it anymore due to his/her better clinical conditions, or because there is a need of tracheostomy or because he/she dies. Specifically they will analyze how the endOclear cleaning maneuver affects microbial colonization in the inner layer of the ETT and how this can determine distal airway inoculation and, ultimately, VAP development.

Specific AIM #1: Investigators will test the hypothesis that routine use of endOclear in patients intubated with a silver-coated ETT will reduce ETT microbial colonization.

Specific AIM #2: Investigators will test the hypothesis that keeping ETTs free from microbial colonization will prevent septic inoculation of distal airways

Specific AIM #3: Investigators will test the hypothesis that prevention of ETT biofilm development will reduce drug resistance rates found in ETT and distal airways isolates

The investigators will conduct a randomized clinical trial on 40 patients intubated with silver-coated ETT and randomized to receive standard ETT cleaning vs cleaning with the endOclear device.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Medical, Surgical or Neuro ICU
* Subjects must be enrolled within 24 hours from intubation
* Subjects expected to be intubated for at least 48 hours or longer
* Subjects have been intubated with a silver-coated ETT

Exclusion Criteria:

* Current and past participation in another interventional trial conflicting with the present study
* Pregnant women
* Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kacmarek, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Pirrone M, Imber DA, Marrazzo F, Pinciroli R, Zhang C, Bry L, Delaney ML, Dubois AM, Thomas JG, Nistico L, Melton-Kreft R, Bittner EA, Kacmarek RM, Berra L. Silver-Coated Endotracheal Tubes Cleaned With a Mechanism for Secretion Removal. Respir Care. 2019 Jan;64(1):1-9. doi: 10.4187/respcare.06222. Epub 2018 Sep 4. PMID 30181363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four patients were found ineligible.
Period: Overall Study
Arm/Group | ETT Cleaning Maneuver | Standard of Care
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETT Cleaning Maneuver | Standard of Care | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (4.1) | 61.2 (3.5) | 63.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 13 | 9 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black/African American | 1 | 2 | 3
  White | 14 | 14 | 28
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Endotracheal Tube Colonization
Description: Discarded ETTs will be collected after extubation and sent for quantitative and qualitative microbiological analysis after silver ion inactivation. Qualitative analysis was based on confocal microscopy, we described visually the distribution of microbial colonization. However, we did not report numerical value because the confounding factors (i.e., number and length of devices).
Time Frame: At extubation (an expected average of 7 days)
Measure: Mean (Standard Deviation); unit: Log colony form unit (CFU)/ mL
Arm/Group | ETT Cleaning Maneuver | Standard of Care
Number analyzed (Participants) | 17 | 19
Log colony form unit (CFU)/ mL | 0.9 (1.2) | 1.6 (1.2)

2. Secondary Outcome: Microbiological Colonization of Distal Airways
Description: Investigators will collect data about distal airways samples performed for clinical reasons during the study period and, in addition, investigators will collect a specimen from the distal airways immediately before extubation.
Time Frame: At extubation (An expected average of 7 days)
Measure: Mean (Standard Deviation); unit: Log colony form unit (CFU)/ mL
Arm/Group | ETT Cleaning Maneuver | Standard of Care
Number analyzed (Participants) | 17 | 19
Log colony form unit (CFU)/ mL | 4.2 (3.8) | 4.8 (4.0)

ADVERSE EVENTS:
Arm/Group | ETT Cleaning Maneuver | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes